CLINICAL TRIAL: NCT04265989
Title: A New Classification and Interventional Therapy for Coronary Artery Ectasia
Acronym: NCIPCAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Chao Yang Hospital (Other); Peking University People's Hospital (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Shubin_Qiao, Director,Head of cardiology department, China National Center for Cardiovascular Diseases
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019XK320064
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Ectasia
Keywords: coronary artery ectasia; new classification; interventional therapy; coronary artery aneurysm
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- coronary artery aneurysm with branches (Experimental): The diameter of coronary artery aneurysm is more than 5mm and less than 10mm, accompany with branches origin from the aneurysm
  Interventions: Device: Single BMS
- coronary artery aneurysm without branches (Experimental): The diameter of coronary artery aneurysm is more than 5mm and less than 10mm, without any branch origin from the aneurysm
  Interventions: Device: Single or Double BMS
- Coronary artery aneurysm with localized stenosis (Experimental): The diameter of coronary artery aneurysm is more than 5mm and less than 10mm, associated with severe stenosis of adjacent sites. localized stenosis defined as lesion to more than 70% stenosis and length less than 20 mm
  Interventions: Device: Single or Double BMS
- Coronary artery aneurysm with diffuse stenosis (Experimental): The diameter of coronary artery aneurysm is more than 5mm and less than 10mm, associated with severe stenosis of adjacent sites. Diffuse stenosis defined as lesion to more than 70% and length more than 20 mm
  Interventions: Device: BMS+DES

INTERVENTIONS:
Device: Single BMS — Single bare metal stent covered the coronary artery aneurysm
  Arms: coronary artery aneurysm with branches
Device: Single or Double BMS — Single or double layer bare metal stents covered the coronary artery aneurysm
  Arms: coronary artery aneurysm without branches
Device: Single or Double BMS — Treated with single or double layer bare metal stents
  Arms: Coronary artery aneurysm with localized stenosis
Device: BMS+DES — Treated with bare metal stent combined with drug eluting stent
  Arms: Coronary artery aneurysm with diffuse stenosis

SUMMARY:
This study is aim to present a new classification for coronary artery ectasia and find the best interventional therapy for different types of patients were treated and studied.

DETAILED DESCRIPTION:
Coronary artery ectasia refers to a variety of reasons cause coronary artery expansion, its diameter is more than 1.5 times that of the adjacent normal coronary artery. Clinical symptoms include angina, myocardial infarction and sudden death.At present, there is no consensus on the mechanism and treatment of the disease, which may be related to the structural failure of the vessel wall and abnormal hemodynamics in the dilated segment.Most of the existing studies are case reports or single-center retrospective analysis of small samples, with low level of evidence.As a common fluid analysis method in the field of engineering, computational fluid dynamics can effectively simulate the movement and stress state of blood under reasonable model assumptions.By comparing the preoperative and postoperative data of real cases, the validity of simulation analysis results can be tested.The purpose of this study is to carry out a multi-center study combining morphological and hemodynamic factors, to propose a new classification and interventional treatment strategy for atherosclerotic coronary artery ectasia, and to provide evidence-based medical evidence for the development of treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged ≥18 years;
* Coronary artery ectasia was confirmed by coronary CT or coronary angiography;
* The patient (or guardian) is fully aware of the study process and signs the informed consent;
* Patients were able to undergo subsequent follow-up.

Exclusion Criteria:

* Congenital coronary artery fistula;
* kawasaki disease;
* Treponema pallidum or lyme treponema;
* Marfan;
* Primary lymphoma;
* Coronary artery pseudoaneurysm;
* Acute infectious disease or autoimmune disease;
* Hematological Disease;
* Severe liver and kidney dysfunction (AMI one week later, alanine transaminase ≥3 times the upper limit of normal value; Creatinine clearance rate ≤30ml/min or blood creatinine ≥2.5mg/dl);
* Unstable craniocerebral disease;
* Cancer;
* Severe cognitive impairment (dementia or severe mental illness);
* Patients with severe physical disabilities who cannot be followed up regularly;
* Other serious uncontrolled systemic diseases;
* Female patient who is ready to become pregnant, already pregnant or nursing;
* Contraindications to percutaneous coronary intervention (PCI) : for patients at high risk of massive bleeding in the digestive tract, intracranial and other areas, or allergic to contrast agents;
* Cannot tolerate dual antiplatelet therapy for at least 1 year;
* Age < 18 years old;
* Patients who are unable or unwilling to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events (MACCEs) | 6 months after treatment
  Number of participants with a composite of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke or urgent target vessel revascularization

SECONDARY OUTCOMES:
Changes in CCS grade | 6 months after treatment
  Number of participants with CCS angina pectoris grade aggravated or alleviate
Changes in drug use | 6 months after treatment
  Number of participants with increased the type or dose of anti-myocardial ischemia drugs
Changes in coronary artery aneurysm diameter | 6 months after treatment
  Number of participants with coronary artery aneurysm diameter reduced, increased or unchanged

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, MD,PhD, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China